CLINICAL TRIAL: NCT06704763
Title: A Drug-Drug Interaction, Single-arm, Open-label Study to Assess the Effect of Quinidine on the Pharmacokinetics of Orforglipron in Healthy Participants
Brief Title: A Drug-Drug Interaction Study of Orforglipron (LY3502970) With Quinidine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 27312; J2A-MC-GZPP (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron; Midazolam; Quinidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Orforglipron (Experimental): Orforglipron administered orally either alone or with another investigational agent
  Interventions: Drug: Orforglipron; Drug: Midazolam; Drug: Quinidine

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
Drug: Midazolam — Administered orally
Drug: Quinidine — Administered orally

SUMMARY:
The purpose of this study is to determine the effect of quinidine on the levels of orforglipron in the blood stream and how long it takes the body to eliminate it, when administered orally in healthy participants.

The study will last up to approximately 8 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG)
* Have a hemoglobin level of:

  * at least 11.4 grams per deciliter (g/dL) for individuals assigned female at birth (AFAB), and
  * at least 12.5 g/dL for individuals assigned male at birth (AMAB)
* Have a body weight equal to or greater than 45 kilograms (kg), and a body mass index within the range of 18.5 to 35.0 kilogram per square meter (kg/m²) at screening

Exclusion Criteria:

* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, psychological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting risk when taking orforglipron, midazolam, or quinidine; or interfering with the interpretation of data
* Have a 12 lead electrocardiogram (ECG) abnormality, including known prolongation of QT/QTc interval, significant bradycardia, significant heart blocks or a history of any risk factors for ventricular arrhythmia, heart failure, hypokalemia or hypomagnesemia, or other factors that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure or pulse rate, deemed to be clinically significant by the investigator
* Have a history of benign ethnic neutropenia
* Have a GI disease or disorder, such as relevant esophageal reflux or gall bladder disease, which could be aggravated by glucagon-like peptide-1 (GLP-1) analogs or impacts gastric emptying, for example gastric bypass surgery or pyloric stenosis, except for appendectomy
* Have a history or presence of pancreatitis, including chronic pancreatitis or idiopathic acute pancreatitis
* Have known allergies to:

  * quinidine
  * midazolam
  * orforglipron
  * related compounds, or
  * any components of the formulation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of Orforglipron | Baseline to Study Completion (Up to 2 Weeks)
  PK: AUC of Orforglipron
PK: Maximum Concentration (Cmax) of Orforglipron | Baseline to Study Completion (Up to 2 Weeks)
  PK: Cmax of Orforglipron

SECONDARY OUTCOMES:
PK: AUC of Midazolam | Baseline to Study Completion (Up to 2 Weeks)
  PK: AUC of Midazolam
PK: Cmax of Midazolam | Baseline to Study Completion (Up to 2 Weeks)
  PK: Cmax of Midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Contact Lilly at 1-800-LillyRx (1-800-545-5979), Study Director — Eli Lilly and Company
Locations (1):
- ICON, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No